CLINICAL TRIAL: NCT05583773
Title: Effects of "ShengXian-QuYu Decoction" on Quality of Life, Symptoms, and Biomarkers in Heart Failure Patients With Reduced and Mildly Reduced Ejection Fraction: a Pragmatic, Nationwide, Multicenter, Parallel Group, Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: SHengXIaN-QuYu DEcoction in Heart Failure With Reduced and Mildly Reduced Ejection Fraction
Acronym: SHINE-HF
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Jingyi Ren, Professor, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-NHLHCRF-LX-02-0102
Record Dates: First submitted 2022-10-08; First posted 2022-10-18 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure
Keywords: ShengXian-QuYu Decoction; Heart failure with reduced ejection fraction; Heart failure with mildly reduced ejection fraction; Quality of life
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ShengXian-QuYu Decoction (Active Comparator): Patients will be randomized 1:1 to either ShengXian-QuYu Decoction or placebo. "ShengXian-QuYu Decoction" (calculated by a medicine): 30g of Astragalus membranaceus (Huangqi), 12g of Cornus officinalis (Shanzhuyu), 9g of Panax ginseng (Hongshen), 12g of Anemarrhena asphodeloides (Zhimu), 8g of Cimicifuga foetida (Shengma), 8g of Bupleurum chinense (Chaihu), 10g of Platycodon grandiflorum (Jiegeng), 10g of Sparganium stoloniferum (Sanleng), 9g of Curcuma phaeocaulis (Ezhu), 3g of Whitmania pigra (Shuizhi).
  Interventions: Drug: ShengXian-QuYu Decoction
- placebo (Placebo Comparator): Placebo matching ShengXian-QuYu Decoction
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ShengXian-QuYu Decoction — Specification: 30ml/bag, given twice daily, per oral use.
  Arms: ShengXian-QuYu Decoction
Other: Placebo — Placebo matching ShengXian-QuYu Decoction, 30ml/bag, given twice daily, per oral use.
  Arms: placebo

SUMMARY:
The purpose of this study is to conduct a multicenter, randomized clinical trial to evaluate the effect of "ShengXian-QuYu Decoction" on quality of life , symptoms, and biomarkers in heart failure patients with reduced and mildly reduced ejection fraction.

DETAILED DESCRIPTION:
This is a pragmatic, nationwide, multicenter, parallel group, randomized, double-blind, placebo-controlled study in patients with heart failure with reduced and mildly ejection fraction, evaluating the effect of "ShengXian-QuYu Decoction" versus placebo, given twice daily in addition to background regional standard of care. The effect of "ShengXian-QuYu Decoction"on quality of life, symptoms and biomarkers will be evaluated.

The primary and secondary endpoints will be examined in subgroups determined by baseline variables reflecting demography, heart failure characteristics, Traditional Chinese Medicine syndrome type, diabetes status, kidney function, left ventricular ejection fraction, natriuretic peptide, and additional co-morbidities, concomitant medications, and others.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥18 years at the time of consent.
2. Established documented diagnosis of symptomatic HFrEF (NYHA functional class II-IV).
3. LVEF <50%.
4. NT-proBNP >600 pg/ml or BNP ≥150 pg/ml (or if hospitalized for heart failure within the previous 12 months, NT-proBNP ≥400 pg/ml or BNP ≥100 pg/ml) at enrolment.
5. Provision of signed informed consent prior to any study specific procedures.

Exclusion Criteria:

1. Current acute decompensated HF or hospitalization due to decompensated HF, ACS, stroke or transient ischemic attack (TIA), coronary revascularization (percutaneous coronary intervention [PCI] or coronary artery bypass grafting [CABG]) or valvular repair/replacement, or other major cardiovascular surgery within 4 weeks prior to enrolment.
2. Uncontrolled severe arrhythmia.
3. Planned to undergo heart transplantation or device implantation.
4. Hepatic impairment aspartate transaminase [AST] or alanine transaminase [ALT] >3x the upper limit of normal [ULN]; or total bilirubin >2x ULN at time of enrolment).
5. Severe infection.
6. eGFR <30 mL/min/1.73 m^2 by CKD-EPI.
7. Active malignancy requiring treatment at the time of visit 1.
8. Women of child-bearing potential who are not willing to use a medically accepted method of contraception that is considered reliable in the judgment of the investigator OR women who have a positive pregnancy test at enrolment or randomization OR women who are breast-feeding.
9. Any condition outside the CV and renal disease area, such as but not limited to malignancy, with a life expectancy of less than 1 years based on investigator's clinical judgement.
10. Systolic blood pressure < 90 mmHg, or systolic blood pressure ≥ 180 mmHg, or diastolic blood pressure ≥ 110 mmHg on 2 consecutive measurements.
11. Heart failure due to infiltrative cardiomyopathies(cardiac amyloidosis, etc.), fulminant myocarditis, constrictive pericarditis.
12. Participation in another clinical study.
13. Inability of the patient, in the opinion of the investigator, to understand and/or comply with study medications, procedures and/or follow-up OR any conditions that, in the opinion of the investigator, may render the patient unable to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2023-03-29 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in the KCCQ Clinical Summary Score | Up to 12 weeks
  KCCQ was a 23-item, self-administered questionnaire that measure the participant's perception of their health status, including their heart failure (HF) symptoms, impact on physical and social function and how their HF impacts the quality of life. KCCQ quantifies 7 domains: physical limitations (6 items), symptom stability (1 item), symptom frequency (4 items), symptom burden (3 items), self-efficacy (2 items), quality of life (3 items) and social limitations (4 items). Scores were generated for each domain and scaled from 0 to 100, with 0 denoting the worst and 100 the best possible status. KCCQ-clinical summary score was average of domains- physical limitation and total symptoms (average of symptom frequency and symptom burden), and transformed to a single score which ranged from 0 (worst) -100 (the best possible status), where the higher score reflected better health status.

SECONDARY OUTCOMES:
Change From Baseline in the Traditional Chinese Medicine Syndrome Score Scale (TCMSSS) | Up to 12 weeks
  Traditional Chinese Medicine Syndrome Score is a instrument that quantifies symptoms. Lower TCM scores reflect better health status.
Change in Exercise Capacity as Measured by the 6-Minutes-Walking-Test (6MWT) Distance | Up to 12 weeks
  Change from baseline to week 12 in exercise capacity as measured by the distance walked in 6 minutes in standardised conditions. Change from baseline was defined as the distance walked in 6 minutes at week 12 minus the baseline value. Baseline value was defined as the last available measurement before start of treatment with randomised study medication.
Change in N-terminal Pro-brain Natriuretic Peptide (NT-proBNP) | Up to 12 weeks
  Change from baseline to week 12 in N-terminal pro-brain natriuretic peptide (NT-proBNP). Baseline value was defined as the mean of all available measurements from the screening visit until start of treatment with randomised study medication.
Change in Left Ventricular Systolic Function | Up to 12 weeks
  Change in left ventricular ejection fraction is assessed by two-dimensional directed M-mode echocardiography.
Change in Left Ventricular End-Diastolic Diameter | Up to 12 weeks
  Change in left ventricular end-diastolic diameter is assessed by two-dimensional directed M-mode echocardiography.
Change in Left Ventricular End-Systolic Diameter | Up to 12 weeks
  Change in left ventricular end-systolic diameter is assessed by two-dimensional directed M-mode echocardiography.
Change in Estimated Glomerular Filtration Rate from Baseline | Up to 12 weeks
  Estimated glomerular filtration rate (eGFR) is calculated by the CKD-EPI equation.
Change From Baseline in the KCCQ Clinical Summary Score | Up to 26 weeks
  KCCQ was a 23-item, self-administered questionnaire that measure the participant's perception of their health status, including their heart failure (HF) symptoms, impact on physical and social function and how their HF impacts the quality of life. KCCQ quantifies 7 domains: physical limitations (6 items), symptom stability (1 item), symptom frequency (4 items), symptom burden (3 items), self-efficacy (2 items), quality of life (3 items) and social limitations (4 items). Scores were generated for each domain and scaled from 0 to 100, with 0 denoting the worst and 100 the best possible status. KCCQ-clinical summary score was average of domains- physical limitation and total symptoms (average of symptom frequency and symptom burden), and transformed to a single score which ranged from 0 (worst) -100 (the best possible status), where the higher score reflected better health status.
Change From Baseline in the Traditional Chinese Medicine Syndrome Score Scale (TCMSSS) | Up to 26 weeks
  Traditional Chinese Medicine Syndrome Score is a instrument that quantifies symptoms. Lower TCM scores reflect better health status.

OTHER OUTCOMES:
Subjects Included in the Composite Endpoint of Cardiovascular Death and Worsening Heart Failure | Up to 12 weeks
  The composite CV endpoint is defined as cardiovascular death, hospitalization due to heart failure or urgent visit required intravenous treatment due to heart failure.
Subjects Included in the Composite Endpoint of Cardiovascular Death and Worsening Heart Failure | Up to 26 weeks
  The composite CV endpoint is defined as cardiovascular death, hospitalization due to heart failure or urgent visit required intravenous treatment due to heart failure.
Renal Composite Endpoint | Up to 12 weeks
  The renal composite endpoint included composite of doubling of serum creatinine (DoSC), end-stage kidney disease (ESKD), and renal death. DoSC: from the baseline average determination (sustained and confirmed by repeat central laboratory measure after at least 30 days and preferably within 60 days). ESKD: initiation of maintenance dialysis for at least 30 days, or renal transplantation, or an eGFR value of <15 mL/min/1.73 m^2 (sustained and confirmed by repeat central laboratory measure after at least 30 days and preferably within 60 days). Renal death: death in participants who have reached ESKD, died without initiating renal replacement therapy, and no other cause of death was determined via adjudication. Adjudication of these events by the EAC was performed in a blinded fashion. Event rate estimated based on the time to the first occurrence of the renal composite endpoint are presented.
Renal Composite Endpoint | Up to 26 weeks
  The renal composite endpoint included composite of doubling of serum creatinine (DoSC), end-stage kidney disease (ESKD), and renal death. DoSC: from the baseline average determination (sustained and confirmed by repeat central laboratory measure after at least 30 days and preferably within 60 days). ESKD: initiation of maintenance dialysis for at least 30 days, or renal transplantation, or an eGFR value of <15 mL/min/1.73 m^2 (sustained and confirmed by repeat central laboratory measure after at least 30 days and preferably within 60 days). Renal death: death in participants who have reached ESKD, died without initiating renal replacement therapy, and no other cause of death was determined via adjudication. Adjudication of these events by the EAC was performed in a blinded fashion. Event rate estimated based on the time to the first occurrence of the renal composite endpoint are presented.
Liver Injury | Up to 12 weeks
  Liver injury is defined as: i) a rise of alanine aminotransferase (ALT) or aspartate aminotransferase (AST) to 3 times above the upper limit of normal [ULN], or ii) a rise of total bilirubin to 2 times above the upper limit of normal [ULN].
Liver Injury | Up to 26 weeks
  Liver injury is defined as: i) a rise of alanine aminotransferase (ALT) or aspartate aminotransferase (AST) to 3 times above the upper limit of normal [ULN], or ii) a rise of total bilirubin to 2 times above the upper limit of normal [ULN].
Bleeding Events | Up to 12 weeks
  All bleeding events, including major bleeding, non-major clinically relevant bleeding and minimal bleeding (for incidences only) will be assessed.
Bleeding Events | Up to 26 weeks
  All bleeding events, including major bleeding, non-major clinically relevant bleeding and minimal bleeding (for incidences only) will be assessed.

CONTACTS AND LOCATIONS:
Locations (26):
- China (26):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing Fengtai Hospital of Integrated Traditional Chinese and Western Medicine, Beijing, Beijing Municipality
  - Dongcheng District First People's Hospital, Beijing, Beijing Municipality
  - Dongfang Hospital Affiliated to Beijing University of Chinese Medicine, Beijing, Beijing Municipality
  - Huairou District Traditional Chinese Medicine Hospital of Beijing, Beijing, Beijing Municipality
  - Beijing Changping Nankou Hospital, Beijing, Beijing Municipality
  - Changping District Traditional Chinese Medicine Hospital, Beijing, Beijing Municipality
  - Tang County Hospital of Traditional Chinese Medicine, Baoding, Hebei
  - Funing Hospital of Traditional Chinese Medicine, Qinhuangdao, Hebei
  - Gongyi City Public Hospital of TCM, Gongyi, Henan
  - Yangzhou Hospital of Traditional Chinese Medicine, Yangzhou, Jiangsu
  - Jining Hospital of Traditional Chinese Medicine, Jining, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - The Affiliated Hospital of Changzhi Institute of Traditional Chinese Medicine, Changzhi, Shanxi
  - Changzhi Medical College Affiliated Heji Hospital, Changzhi, Shanxi
  - Changzhi Hospital of Traditional Chinese Medicine, Changzhi, Shanxi
  - Chengdu Integrated TCM and Western Medicine Hospital, Chengdu, Sichuan
  - Jixian Chinese Traditional Hospital, Tianjin, Tianjin Municipality
  - Urumqi Hospital of Traditional Chinese Medicine, Ürümqi, Xinjiang
  - Korla Hospital of Traditional Chinese Medicine, Bayan Gol Autonomous Prefecture, Xinjiang Uygur Autonomous Region
  - Changji Hospital of Traditional Chinese Medicine, Changji Hui Autonomous Prefecture, Xinjiang Uygur Autonomous Region
  - Gulja Hospital of Traditional Chinese Medicine, Ili Kazakh Autonomous Prefecture, Xinjiang Uygur Autonomous Region
  - Zhaosu Hospital of Traditional Chinese Medicine, Ili Kazakh Autonomous Prefecture, Xinjiang Uygur Autonomous Region
  - Xinyuan Traditional Chinese Medicine Hospital, Ili Kazakh Autonomous Prefecture, Xinjiang Uygur Autonomous Region
  - Linhai Hospital of Traditional Chinese Medicine, Linhai, Zhejiang

IPD SHARING:
Plan to Share IPD: No